CLINICAL TRIAL: NCT01712750
Title: Near-Infrared Spectroscopic (NIRS) Tissue Oxygen Saturation and the Vascular Occlusion Test in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre (Other)
Other Study IDs: REB-17456
Record Dates: First submitted 2012-10-23; First posted 2012-10-24 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Vascular Occlusion Test
Keywords: Regional tissue oximetry; Cardiopulmonary bypass; Cardiac surgical procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VOT on bypass

SUMMARY:
Tissue oxygen saturation (StO2) and its recovery during a vascular occlusion test (VOT) will be measured in elective cardiac surgery patients undergoing cardiopulmonary bypass using a non-invasive near infrared spectrometry (NIRS) machine. The purpose of this study is to determine whether changes in VOT measurements occur in patients during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult, elective cardiac surgery patients
* Procedure using cardiopulmonary bypass

Exclusion Criteria:

* Contraindication to pneumatic cuff inflation
* Pregnant
* Significant peripheral vascular disease of the arms
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective cardiac surgery patients undergoing coronary artery bypass and valve surgery using cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-02; Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
VOT reperfusion slope | Intra-operative (within 12 hours)
  Reperfusion slope as measured during vascular occlusion test in units of %/s

CONTACTS AND LOCATIONS:
Overall Officials: John M Murkin, MD, FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada